CLINICAL TRIAL: NCT01162564
Title: Single-Arm, Prospective, Multi-Center Observational Study of a Flexible Composite Next Generation Tissue Separating Mesh(NG-TSM)to Assess Ease of Use and Early Outcomes in Laparoscopic Incisional/Ventral Hernia
Brief Title: Flexible Composite Next Generation Tissue Separating Mesh in Laparoscopic Incisional/Ventral Hernia Repair
Status: Completed | Type: Observational
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Lynn McRoy MD / Medical Director, Ethicon
Other Study IDs: 200-10-002
Record Dates: First submitted 2010-07-13; First posted 2010-07-14 (Estimated); Last update posted 2011-04-27 (Estimated); Status verified 2011-04

CONDITIONS: Incisional Hernia; Ventral Hernia
MeSH Terms: conditions — Incisional Hernia; Hernia, Ventral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NG-TSM: Patients receiving NG-TSM to repair an abdominal incisional/ventral hernia
  Interventions: Device: NG-TSM

INTERVENTIONS:
Device: NG-TSM — Flexible Composite Next Generation Tissue Separating Mesh
  Other Names: Ethicon Physiomesh

SUMMARY:
This is a multi-center, observational study of incisional/ventral hernia repair with NG-TSM laparoscopically. The study is not randomized and has a single treatment design assessing NG-TSM intra-operatively, its ease of use and handling characteristics.

DETAILED DESCRIPTION:
The objectives of the study are to evaluate the ease of use of NG-TSM intra-operatively in laparoscopic incisional/ventral hernia repair, and assessing early outcomes post-operatively following mesh implantation, including seroma formation, hematoma, wound complications, infections, early recurrences, adverse events, and subject comfort, as well as health economic data to include quality of life, subject satisfaction data, time of procedure, length of stay, re-hospitalization, and extended hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be able to provide written informed consent
* Male or female subjects that are ≥ 18 years of age
* Female subjects must be using adequate contraception, or be surgically sterile, postmenopausal or practicing abstinence, and not planning to become pregnant
* Planned laparoscopic procedure to repair an abdominal incisional/ventral hernia that requires the addition of reinforcing or bridging material to obtain the desired surgical result

Exclusion Criteria:

* Subjects with a potential growth as NGTSM will not stretch significantly
* Female subjects who are pregnant on the day of implantation
* Surgical site (mesh implantation site) that is classified as contaminated (acute, non purulent, inflamed) or dirty/infected (containing retained devitalized tissue and those that involve existing clinical infection or perforated viscera)
* Subjects who have received investigational articles less than 30 days prior to enrollment or who are currently receiving investigational products or devices
* Employees of the investigator or study center with direct involvement in the proposed study or other studies under the direction of that investigator or study center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for planned laparoscopic procedure to repair an abdominal incisional/ventral hernia that requires the addition of reinforcing or bridging material to obtain the desired surgical result
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2010-06; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn McRoy, MD, Study Director — Ethicon, Inc.
Locations (6):
- United States (6):
  - Capital Region Hospital, Jefferson City, Missouri
  - Washington University School of Medicine / Dept of Surgery, St Louis, Missouri
  - Montefiore Medical Center, The Bronx, New York
  - First Health Moore Regional Hospital, Pinehurst, North Carolina
  - New Hanover Regional Hospital, Wilmington, North Carolina
  - Eastern Virginia Medical School, Norfolk, Virginia